CLINICAL TRIAL: NCT03495492
Title: Dermal Chelation Lowers White Blood Cell Count in Chronic Lymphocytic Leukemia
Brief Title: Chronic Lymphocytic Leukemia Responds to Dermal Chelation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Optimum Health, Natural Healthcare Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCCLL2018
Record Dates: First submitted 2018-02-14; First posted 2018-04-12 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; CLL; Dermal Chelation; Nutritional Therapy
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Nutrition Therapy

STUDY DESIGN:
Intervention Model Description: Clinical trials with a single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants (Experimental): Group receiving dermal chelation and nutritional therapy
  Interventions: Device: Dermal Chelation; Dietary Supplement: Nutritional Therapy

INTERVENTIONS:
Device: Dermal Chelation — Dermal chelation with Aqua DetoxTM system for one or more hours one or more times each week.
Dietary Supplement: Nutritional Therapy — Vitamins and minerals that will be taken one or more times a day.

SUMMARY:
The purpose of this clinical trial is to identify 50 participants with Chronic Lymphocytic Leukemia (CLL) and follow their total white blood cell (WBC) counts and absolute lymphocyte counts after performing dermal chelation and administering nutritional therapy

DETAILED DESCRIPTION:
The purpose of this clinical trial is to use dermal chelation and hair tissue analysis to identify 50 participants with CLL. The total wbc counts and absolute lymphocyte counts of these participants will be followed after serial dermal chelations and nutritional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Chronic Lymphocytic Leukemia and has a toxic heavy metal load
* Toxic heavy metal load

Exclusion Criteria:

* Pregnant
* Pacemaker implants
* Organ transplant recipients
* Psychotic episodes or epileptic seizures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Serial Total White Blood Cell Count | up to 12 months
  Total WBC counts taken on a regular interval.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Richter PA, Bishop EE, Wang J, Swahn MH. Tobacco smoke exposure and levels of urinary metals in the U.S. youth and adult population: the National Health and Nutrition Examination Survey (NHANES) 1999-2004. Int J Environ Res Public Health. 2009 Jul;6(7):1930-46. doi: 10.3390/ijerph6071930. Epub 2009 Jul 2. PMID 19742163
- [Result] Sandborgh-Englund G, Elinder CG, Johanson G, Lind B, Skare I, Ekstrand J. The absorption, blood levels, and excretion of mercury after a single dose of mercury vapor in humans. Toxicol Appl Pharmacol. 1998 May;150(1):146-53. doi: 10.1006/taap.1998.8400. PMID 9630463
- [Result] Yaginuma-Sakurai K, Murata K, Iwai-Shimada M, Nakai K, Kurokawa N, Tatsuta N, Satoh H. Hair-to-blood ratio and biological half-life of mercury: experimental study of methylmercury exposure through fish consumption in humans. J Toxicol Sci. 2012 Feb;37(1):123-30. doi: 10.2131/jts.37.123. PMID 22293416
- [Result] Tchounwou PB, Yedjou CG, Patlolla AK, Sutton DJ. Heavy metal toxicity and the environment. Exp Suppl. 2012;101:133-64. doi: 10.1007/978-3-7643-8340-4_6. PMID 22945569
- [Result] Barry PS. A comparison of concentrations of lead in human tissues. Br J Ind Med. 1975 May;32(2):119-39. doi: 10.1136/oem.32.2.119. PMID 1131339
- [Result] Vaglenov A, Creus A, Laltchev S, Petkova V, Pavlova S, Marcos R. Occupational exposure to lead and induction of genetic damage. Environ Health Perspect. 2001 Mar;109(3):295-8. doi: 10.1289/ehp.01109295. PMID 11333192
- [Result] Wani AL, Ara A, Usmani JA. Lead toxicity: a review. Interdiscip Toxicol. 2015 Jun;8(2):55-64. doi: 10.1515/intox-2015-0009. PMID 27486361
- [Result] Nie LH, Wright RO, Bellinger DC, Hussain J, Amarasiriwardena C, Chettle DR, Pejovic-Milic A, Woolf A, Shannon M. Blood lead levels and cumulative blood lead index (CBLI) as predictors of late neurodevelopment in lead poisoned children. Biomarkers. 2011 Sep;16(6):517-24. doi: 10.3109/1354750X.2011.604133. Epub 2011 Aug 9. PMID 21827276
- [Result] Jo S, Woo HD, Kwon HJ, Oh SY, Park JD, Hong YS, Pyo H, Park KS, Ha M, Kim H, Sohn SJ, Kim YM, Lim JA, Lee SA, Eom SY, Kim BG, Lee KM, Lee JH, Hwang MS, Kim J. Estimation of the Biological Half-Life of Methylmercury Using a Population Toxicokinetic Model. Int J Environ Res Public Health. 2015 Jul 31;12(8):9054-67. doi: 10.3390/ijerph120809054. PMID 26264017
- [Result] Rooney JP. The retention time of inorganic mercury in the brain--a systematic review of the evidence. Toxicol Appl Pharmacol. 2014 Feb 1;274(3):425-35. doi: 10.1016/j.taap.2013.12.011. Epub 2013 Dec 22. PMID 24368178
- [Result] Cretacci Y, Parsons PJ. Localized accumulation of lead within and among bones from lead-dosed goats. Environ Res. 2010 Jan;110(1):26-32. doi: 10.1016/j.envres.2009.09.005. PMID 19897186
- [Result] Flood PR, Schmidt PF, Wesenberg GR, Gadeholt H. The distribution of lead in human hemopoietic tissue and spongy bone after lead poisoning and Ca-EDTA chelation therapy. Observations made by atomic absorption spectroscopy, laser microbeam mass analysis and electron microbeam X-ray analysis. Arch Toxicol. 1988;62(4):295-300. doi: 10.1007/BF00332490. PMID 3149183
- [Result] Stelzer KJ, Pazdernik TL. Cadmium-induced immunotoxicity. Int J Immunopharmacol. 1983;5(6):541-8. doi: 10.1016/0192-0561(83)90047-4. PMID 6363310
- [Result] Bauchinger M, Schmid E, Einbrodt HJ, Dresp J. Chromosome aberrations in lymphocytes after occupational exposure to lead and cadmium. Mutat Res. 1976 Jan;40(1):57-62. doi: 10.1016/0165-1218(76)90023-9. No abstract available. PMID 1250252
- [Result] Grujic S, Ristic M, Lausevic M. Heavy metals in petroleum-contaminated surface soils in Serbia. Ann Chim. 2004 Dec;94(12):961-70. doi: 10.1002/adic.200490118. PMID 15689032
- [Result] Stigter JB, de Haan HP, Guicherit R, Dekkers CP, Daane ML. Determination of cadmium, zinc, copper, chromium and arsenic in crude oil cargoes. Environ Pollut. 2000 Mar;107(3):451-64. doi: 10.1016/s0269-7491(99)00123-2. PMID 15092991
- [Result] Cline DM, Hiott DW, Nunnery KE, Shealy RG, Towles WC, Watkins RW. Pneumatosis cystoides intestinalis. J S C Med Assoc. 1973 Jun;69(6):226-8. No abstract available. PMID 4513535
- [Result] Kang Y, Larson SB, Robins RK, Revankar GR. Synthesis and biological evaluation of certain 3-beta-D-ribofuranosyl-1,2,4-triazolo[4,3-b)pyridazines related to formycin prepared via ring closure of pyridazine precursors. J Med Chem. 1989 Jul;32(7):1547-51. doi: 10.1021/jm00127a024. PMID 2738890
- [Result] Farooqui AA, Roy AB. The sulphatase of ox liver. XX. The preparation of sulphatases B1alpha and B1beta. Biochim Biophys Acta. 1976 Dec 8;452(2):431-9. doi: 10.1016/0005-2744(76)90193-5. PMID 1009120
- [Result] Van Neste D. Why care about linear hair growth rates (LHGR)? a study using in vivo imaging and computer assisted image analysis after manual processing (CAIAMP) in unaffected male controls and men with male pattern hair loss (MPHL). Eur J Dermatol. 2014 Sep-Oct;24(5):568-76. doi: 10.1684/ejd.2014.2428. PMID 25445091
- [Result] Van Neste D. Thickness, medullation and growth rate of female scalp hair are subject to significant variation according to pigmentation and scalp location during ageing. Eur J Dermatol. 2004 Jan-Feb;14(1):28-32. PMID 14965792
- [Result] Li J, Cen D, Huang D, Li X, Xu J, Fu S, Cai R, Wu X, Tang M, Sun Y, Zhang J, Zheng J. Detection and analysis of 12 heavy metals in blood and hair sample from a general population of Pearl River Delta area. Cell Biochem Biophys. 2014 Dec;70(3):1663-9. doi: 10.1007/s12013-014-0110-6. PMID 25009099
- [Result] Vorob'ev VI, Kosjuk GN. Distribution of repetitive and non-repetitive nucleotide sequences in the DNA of sea urchin. FEBS Lett. 1974 Oct 1;47(1):43-6. doi: 10.1016/0014-5793(74)80422-9. No abstract available. PMID 4609793
- [Result] McCabe MJ Jr, Lawrence DA. Lead, a major environmental pollutant, is immunomodulatory by its differential effects on CD4+ T cells subsets. Toxicol Appl Pharmacol. 1991 Oct;111(1):13-23. doi: 10.1016/0041-008x(91)90129-3. PMID 1719661
- [Result] Devi KD, Banu BS, Grover P, Jamil K. Genotoxic effect of lead nitrate on mice using SCGE (comet assay). Toxicology. 2000 Apr 14;145(2-3):195-201. doi: 10.1016/s0300-483x(00)00154-2. PMID 10771143
- [Result] Bernhoft RA. Mercury toxicity and treatment: a review of the literature. J Environ Public Health. 2012;2012:460508. doi: 10.1155/2012/460508. Epub 2011 Dec 22. PMID 22235210
- [Result] Rose TP. Sterilization of carious dentine with silver nitrate. Chronicle. 1976 Oct;39(8):151, 159. No abstract available. PMID 1068773
- [Result] Vainio H, Sorsa M. Chromosome aberrations and their relevance to metal carcinogenesis. Environ Health Perspect. 1981 Aug;40:173-80. doi: 10.1289/ehp.8140173. PMID 7023931
- [Result] Bass DA, Hickock D, Quig D, Urek K. Trace element analysis in hair: factors determining accuracy, precision, and reliability. Altern Med Rev. 2001 Oct;6(5):472-81. PMID 11703167
- [Result] Niculescu T, Dumitru R, Botha V, Alexandrescu R, Manolescu N. Relationship between the lead concentration in hair and occupational exposure. Br J Ind Med. 1983 Feb;40(1):67-70. doi: 10.1136/oem.40.1.67. PMID 6824602
- [Result] Mohamed Fel B, Zaky EA, El-Sayed AB, Elhossieny RM, Zahra SS, Salah Eldin W, Youssef WY, Khaled RA, Youssef AM. Assessment of Hair Aluminum, Lead, and Mercury in a Sample of Autistic Egyptian Children: Environmental Risk Factors of Heavy Metals in Autism. Behav Neurol. 2015;2015:545674. doi: 10.1155/2015/545674. Epub 2015 Oct 5. PMID 26508811
- [Result] Jung SY, Kim S, Lee K, Kim JY, Bae WK, Lee K, Han JS, Kim S. Association between secondhand smoke exposure and blood lead and cadmium concentration in community dwelling women: the fifth Korea National Health and Nutrition Examination Survey (2010-2012). BMJ Open. 2015 Jul 16;5(7):e008218. doi: 10.1136/bmjopen-2015-008218. PMID 26185180
- [Result] Horiguchi H, Oguma E, Kayama F. Cadmium induces anemia through interdependent progress of hemolysis, body iron accumulation, and insufficient erythropoietin production in rats. Toxicol Sci. 2011 Jul;122(1):198-210. doi: 10.1093/toxsci/kfr100. Epub 2011 May 3. PMID 21540277
- See also: Mercury section in Chapter 33 — https://booksite.elsevier.com/samplechapters/9780123694133/Sample_Chapters/01~Front_Matter.pdf
- See also: National Institute of Environmental Health Science Information on Mercury — https://www.niehs.nih.gov/health/topics/agents/mercury/index.cfm
- See also: Mayo Clinic. "Enlarged spleen (splenomegaly)." Mayo Foundation for Medical Education and Research (MFMER) 1998-2017. — https://www.mayoclinic.org/diseases-conditions/enlarged-spleen/symptoms-causes/syc-20354326
- See also: Jacob, Harry S. "Overview of the spleen." Merck Manual. Last full review/revision November 2016 — http://www.merckmanuals.com/home/blood-disorders/spleen-disorders/overview-of-the-spleen
- See also: American Cancer Society. What Is Acute Lymphocytic Leukemia? The American Cancer Society medical and editorial content team. Last Medical Review: December 2, 2014 Last Revised: February 18, 2016. — https://www.cancer.org/cancer/acute-lymphocytic-leukemia/about/what-is-all.html
- See also: Chapter 153, The White Blood Cell and Differential Count — https://www.ncbi.nlm.nih.gov/books/NBK261/
- See also: Key Statistics for Chronic Lymphocytic Leukemia — https://www.cancer.org/cancer/chronic-lymphocytic-leukemia/about/key-statistics.html
- See also: Mayo Clinic's Information on Leukemia — https://www.mayoclinic.org/diseases-conditions/leukemia/symptoms-causes/syc-20374373
- See also: Mayo Clinic's Information on Chronic Lymphocytic Leukemia — https://www.mayoclinic.org/diseases-conditions/chronic-lymphocytic-leukemia/diagnosis-treatment/drc-20352433
- See also: Johns Hopkins Medicine. Leukemia Treatments. The Sidney Kimmel Comprehensive Cancer Center — https://www.hopkinsmedicine.org/kimmel_cancer_center/centers/leukemia_program/current_treatments.html
- See also: Liver and Cadmium Toxicity. J Drug Metabol Toxicology — https://www.omicsonline.org/liver-and-cadmium-toxicity-2157-7609.S5-001.php?aid=3686
- See also: New Jersey Department of Health. Right to Know Hazardous Substance Fact Sheet. Revision 4/2010 — http://nj.gov/health/eoh/rtkweb/documents/fs/1349.pdf
- See also: Center for Drug Evaluation and Research. Environmental Assessment and Finding of no Significant Impact of Nicotine Inhaler (Nicotine Inhalation System). Food and Drug Administration. Date completed: 3/5/1977. — https://www.accessdata.fda.gov/drugsatfda_docs/nda/97/20714_NICOTROL%20INHALER%2010MG,%20CARTRIDE_EAFONSI.PDF
- See also: National Cancer Institute. Cancer Stat Facts: Leukemia. Surveillance, Epidemiology, and End Results (SEER) Program of the National Cancer Institute. SEER Data, 1973-2014. — https://seer.cancer.gov/statfacts/html/leuks.html
- See also: National Cancer Institute at the National Institutes of Health. Chronic Lymphocytic Leukemia Treatment. Updated: October 26, 2017. — https://www.cancer.gov/types/leukemia/hp/cll-treatment-pdq#section/_30
- See also: Johns Hopkins Medicine. Leukemia Treatments. The Sidney Kimmel Comprehensive Cancer Center 1973- — https://www.hopkinsmedicine.org/kimmel_cancer_center/centers/leukemia_program/current_treatments.html
- See also: Mayo Clinic. Chronic lymphocytic leukemia. Blood Test Information — https://www.mayoclinic.org/diseases-conditions/chronic-lymphocytic-leukemia/diagnosis-treatment/drc-20352433
- See also: American Society of Clinical Oncology (ASCO). Leukemia - Chronic Lymphocytic - CLL: Statistics. Approved by the Cancer.Net Editorial Board, 06/2016 — https://www.cancer.net/cancer-types/leukemia-chronic-lymphocytic-cll/statistics